CLINICAL TRIAL: NCT01648738
Title: Effectiveness of a Short, Intensive and Standardised Spa Therapy for Subacute and Chronic Low Back Pain on Return to Work for Patients in Sick Leave From 4 to 24 Weeks Duration : a Randomized Controlled Trial Using a Modified Zelen Method
Brief Title: Effectiveness of a Short, Intensive and Standardised Spa Therapy for Low Back Pain on Sick Leave Duration
Acronym: ITILO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/04
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Low Back Pain
Keywords: Subacute low back pain; Chronic low back pain; Low back pain; Disability; Education; Exercise; Spa therapy; Physiotherapy; Multidisciplinary; Cost-effectiveness; Sick leave
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spa therapy, exercise and educational therapy (Experimental): Spa therapy, exercise and educational therapy
  Interventions: Other: Spa therapy, exercise and educational therapy
- Usual care and counselling (Back book) (Active Comparator): Usual care and counselling (Back book)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Spa therapy, exercise and educational therapy — During 5 days: Spa therapy (2 hours/day), exercises (30 min/day), educational therapy (45 min/day) including education on physical activities, work, and pain management
  Other Names: multidisciplinary program
  Arms: Spa therapy, exercise and educational therapy
Other: Usual care — Information, counseling, treatment usually provided for sub-acute and chronic low back pain and the back book
  Arms: Usual care and counselling (Back book)

SUMMARY:
The purpose of this study is to determine whether an intensive 5 days long multidisciplinary program (including spa therapy, exercises and patients'education) is more effective regarding return to work than usual care in subacute and chronic low back pain for people in sick leave from 4 to 24 weeks duration, and for which an extension of sick leave is considered

DETAILED DESCRIPTION:
Sick leave due to low back pain (LBP) is costly and compromises workforce productivity. Sick leave itself, fears and believes regarding return to work, and a low self-esteem have been identified as independent predictors of extended sick leave. Previous data suggested that multidisciplinary rehabilitation programs, including physical activities and psychobehavioral management, should decrease sick leave duration in chronic LBP. However these programs are heavy (at least 4 weeks long), and are often proposed to patients at the end of the management (over 6 months after the beginning of symptoms). Another approach could be to propose a shorter multidisciplinary program (for example 5 days long), earlier in the history of LBP to break the vicious circle as soon as possible. The target population could be people suffering from subacute LBP with sick leave duration between 4 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 60 years (included)
* Low back pain (or back and radicular pain with back pain the most painful)
* Sick leave between 4 and 24 weeks duration, without expected return to work
* A prior medical evaluation is made and the results will be communicated to the patient
* Patient giving his informed consent to participate in the study
* Patient affiliated to or beneficiary of social insurance

Exclusion Criteria:

* Cognition or behavioral disorders making it impossible to assess
* Inability to speak and write French
* Contra-indication to perform a short spa therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Frequency of return to work | 1 year
  Frequency of return to work 1 year after the inclusion date

SECONDARY OUTCOMES:
Pain | Every 2 weeks during 1 year
  Evaluated by the area under the curve of pain (numeric scale from 0 to 100) assessed every 2 weeks during 1 year
Function | 1 year
  Assessed with QUEBEC functional scale
Quality of life | 1 year
  Assessed with MOS SF- 12
TWIST | 1 year
  Time without symptom (without pain)
Sick leave | 1 year
  Number of sick leave days from 6 to 12 months after inclusion date

CONTACTS AND LOCATIONS:
Overall Officials: Serge POIRAUDEAU, MD PhD, Principal Investigator — Cochin Hospital and Descartes University, INSERM; Emmanuel COUDEYRE, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand; Arnaud DUPEYRON, MD, PhD, Principal Investigator — Groupe Hospitalo-Universitaire Carémeau; Ygal ATTAL, MD, Principal Investigator; Jean-Max TESSIER, MD, Principal Investigator — Hôpital Thermal de Dax
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Boutron I, Tubach F, Giraudeau B, Ravaud P. Blinding was judged more difficult to achieve and maintain in nonpharmacologic than pharmacologic trials. J Clin Epidemiol. 2004 Jun;57(6):543-50. doi: 10.1016/j.jclinepi.2003.12.010. PMID 15246122
- [Background] Boutron I, Guittet L, Estellat C, Moher D, Hrobjartsson A, Ravaud P. Reporting methods of blinding in randomized trials assessing nonpharmacological treatments. PLoS Med. 2007 Feb;4(2):e61. doi: 10.1371/journal.pmed.0040061. PMID 17311468
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] Coudeyre E, Tubach F, Rannou F, Baron G, Coriat F, Brin S, Revel M, Poiraudeau S. Effect of a simple information booklet on pain persistence after an acute episode of low back pain: a non-randomized trial in a primary care setting. PLoS One. 2007 Aug 8;2(8):e706. doi: 10.1371/journal.pone.0000706. PMID 17684553
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Druss BG, Rosenheck RA, Sledge WH. Health and disability costs of depressive illness in a major U.S. corporation. Am J Psychiatry. 2000 Aug;157(8):1274-8. doi: 10.1176/appi.ajp.157.8.1274. PMID 10910790
- [Background] Hansson TH, Hansson EK. The effects of common medical interventions on pain, back function, and work resumption in patients with chronic low back pain: A prospective 2-year cohort study in six countries. Spine (Phila Pa 1976). 2000 Dec 1;25(23):3055-64. doi: 10.1097/00007632-200012010-00013. PMID 11145817
- [Background] Magnussen L, Nilsen S, Raheim M. Barriers against returning to work--as perceived by disability pensioners with back pain: a focus group based qualitative study. Disabil Rehabil. 2007 Feb 15;29(3):191-7. doi: 10.1080/09638280600747793. PMID 17364769
- [Background] Costa Lda C, Maher CG, McAuley JH, Hancock MJ, Herbert RD, Refshauge KM, Henschke N. Prognosis for patients with chronic low back pain: inception cohort study. BMJ. 2009 Oct 6;339:b3829. doi: 10.1136/bmj.b3829. PMID 19808766
- [Background] Nguyen M, Revel M, Dougados M. Prolonged effects of 3 week therapy in a spa resort on lumbar spine, knee and hip osteoarthritis: follow-up after 6 months. A randomized controlled trial. Br J Rheumatol. 1997 Jan;36(1):77-81. doi: 10.1093/rheumatology/36.1.77. PMID 9117181
- [Background] Quilty B, Tucker M, Campbell R, Dieppe P. Physiotherapy, including quadriceps exercises and patellar taping, for knee osteoarthritis with predominant patello-femoral joint involvement: randomized controlled trial. J Rheumatol. 2003 Jun;30(6):1311-7. PMID 12784408
- [Background] Poiraudeau S, Rannou F, Le Henanff A, Coudeyre E, Rozenberg S, Huas D, Martineau C, Jolivet-Landreau I, Revel M, Ravaud P. Outcome of subacute low back pain: influence of patients' and rheumatologists' characteristics. Rheumatology (Oxford). 2006 Jun;45(6):718-23. doi: 10.1093/rheumatology/kei231. Epub 2005 Dec 23. PMID 16377729
- [Background] Reme SE, Hagen EM, Eriksen HR. Expectations, perceptions, and physiotherapy predict prolonged sick leave in subacute low back pain. BMC Musculoskelet Disord. 2009 Nov 13;10:139. doi: 10.1186/1471-2474-10-139. PMID 19912626
- [Background] Roberts PJ, Roberts C, Sibbald B, Torgerson DJ. Increasing response rates to postal questionnaires. Effect of incentives on response rates must be considered. BMJ. 2002 Aug 24;325(7361):444. No abstract available. PMID 12201284
- [Background] Savigny P, Watson P, Underwood M; Guideline Development Group. Early management of persistent non-specific low back pain: summary of NICE guidance. BMJ. 2009 Jun 4;338:b1805. doi: 10.1136/bmj.b1805. No abstract available. PMID 19502217
- [Background] Schonstein E, Kenny DT, Keating J, Koes BW. Work conditioning, work hardening and functional restoration for workers with back and neck pain. Cochrane Database Syst Rev. 2003;(1):CD001822. doi: 10.1002/14651858.CD001822. PMID 12535416
- [Background] Waddell G, Burton AK. Occupational health guidelines for the management of low back pain at work: evidence review. Occup Med (Lond). 2001 Mar;51(2):124-35. doi: 10.1093/occmed/51.2.124. PMID 11307688
- [Background] Wood L, Egger M, Gluud LL, Schulz KF, Juni P, Altman DG, Gluud C, Martin RM, Wood AJ, Sterne JA. Empirical evidence of bias in treatment effect estimates in controlled trials with different interventions and outcomes: meta-epidemiological study. BMJ. 2008 Mar 15;336(7644):601-5. doi: 10.1136/bmj.39465.451748.AD. Epub 2008 Mar 3. PMID 18316340
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Karjalainen K, Malmivaara A, van Tulder M, Roine R, Jauhiainen M, Hurri H, Koes B. Multidisciplinary biopsychosocial rehabilitation for subacute low back pain among working age adults. Cochrane Database Syst Rev. 2003;(2):CD002193. doi: 10.1002/14651858.CD002193. PMID 12804427
- [Background] Anema JR, Steenstra IA, Bongers PM, de Vet HC, Knol DL, Loisel P, van Mechelen W. Multidisciplinary rehabilitation for subacute low back pain: graded activity or workplace intervention or both? A randomized controlled trial. Spine (Phila Pa 1976). 2007 Feb 1;32(3):291-8; discussion 299-300. doi: 10.1097/01.brs.0000253604.90039.ad. PMID 17268258
- [Result] Nguyen C, Boutron I, Rein C, Baron G, Sanchez K, Palazzo C, Dupeyron A, Tessier JM, Coudeyre E, Eschalier B, Forestier R, Roques-Latrille CF, Attal Y, Lefevre-Colau MM, Rannou F, Poiraudeau S. Intensive spa and exercise therapy program for returning to work for low back pain patients: a randomized controlled trial. Sci Rep. 2017 Dec 20;7(1):17956. doi: 10.1038/s41598-017-18311-z. PMID 29263353
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29263353